CLINICAL TRIAL: NCT04164797
Title: A Clinical Study of Endostar Combined With TP Regimen for Chemoradiotherapy in Esophageal Cancer
Brief Title: Study of Endostar Combined With TP Regimen for Esophageal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SecondXianJiaotongU
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Patients With Esophageal Cancer(Ⅱ-Ⅲ)
Keywords: endostar Esophageal Cancer
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): endostar : 7.5mg/m2/d,continuous infusion for 5 days in week 1、3、5、7, chemotherapy：paclitaxel liposomes 50mg / m2, ivgtt, d8, 15, 22, 29, 36, carboplatin AUC 2, ivgtt d8, 15, 22, 29, 36 radiotherapy：EBRT，61.2 Gy，1.8Gy/d
  Interventions: Drug: endostar+chemoradiotherapy
- control group (Active Comparator): chemotherapy：paclitaxel liposomes 50mg / m2, ivgtt, d8, 15, 22, 29, 36, carboplatin AUC 2, ivgtt d8, 15, 22, 29, 36 radiotherapy：EBRT，61.2 Gy，1.8Gy/d
  Interventions: Other: chemoradiotherapy

INTERVENTIONS:
Drug: endostar+chemoradiotherapy — antiangiogenic drug+chemoradiotherapy
  Arms: treatment group
Other: chemoradiotherapy — chemoradiotherapy
  Arms: control group

SUMMARY:
a randomized controlled trial of endostar combined with TP regimen(liposomal paclitaxel-carboplatin) for chemoradiotherapy in esophageal squamous cell carcinoma(Ⅱ-Ⅲ)

DETAILED DESCRIPTION:
This study was a controlled clinical trial.A total of 402 patients with pathologically confirmed esophageal squamous cell carcinoma would be enrolled.Patients were randomly divided into two group ,with 201 in the treatment group and 201 in the control group.The treatment group was treated with endostar,chemotherapy (liposomal paclitaxel-carboplatin)and concurrent radiotherapy.The control group was treated with chemotherapy (liposomal paclitaxel-carboplatin)and concurrent radiotherapy .The efficiency and safety would be evaluated. The objective response rate and progress free survival would be analyzed.This data of this study might provide a more effective treatment for esophageal squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years;
2. Pathology confirmed as esophageal squamous cell carcinoma and Clinical stage is II-III;
3. Initial treatment, No surgery history;
4. ECOG 0~2;
5. Expected survival >=3 months;
6. All the patients should have target lesions that are measurable and evaluable;
7. Should be able to consume liquid diet, no esophageal perforation symptoms, no distant metastases;
8. The main organ function is normal, which meets the following criteria:

(1) The standard of blood test should be met (14 days without blood transfusion and blood products, no G-CSF and other hematopoietic stimulation factor correction): Hb>=100g/L;ANC>=1.5x10^9/L;PLT>=100x10^9/L; (2) Biochemical inspection shall meet the following criteria: TBIL < 1.5 ULN; ALT and AST < 2.0 ULN.Serum Cr is less than 1.5 ULN or endogenous creatinine clearance rate > 50 ml/min (the Cockcroft Gault formula); (3) Pulmonary function FEV1 >=1 L or >50% of corresponding value of normal people;

9. Female during the reproductive period should be ensured contraception during the study period; 10. Participants voluntarily joined the study, signed informed consent, and had good compliance and follow-up.

Exclusion Criteria:

1. Patients who do not meet the pathological type of the inclusion criteria and the primary site;
2. Allergic to recombinant endostar, carboplatin, paclitaxel, and contrast agents;
3. Have a distant metastasis;
4. The primary focal tumors or lymph node already had a surgical treatment (except for biopsy), chemoradiotherapy or targeted therapy;
5. Patient who suffered from other malignant tumor;
6. Subject with severe pulmonary and cardiopathic disease history;
7. Pregnant woman or Lactating Women and Women in productive age who refuse take contraception in observation period;
8. Subject with a Personality or psychiatric diseases, people with no legal capacity or people with limited capacity for civil conduct;
9. Received other medicine trials in past 4 weeks;
10. Refuse or incapable to sign the informed consent form of participating this trial;
11. The researchers judged other conditions that could affect clinical research and the results of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2019-11-25 (Estimated); Primary Completion 2021-07-13 (Estimated); Study Completion 2021-07-13 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | Time Frame: approximately 18 months
  complete response(CR)+partial response(PR) according to RECIST 1.1
progression-free survival(PFS) | Time Frame: approximately 36 months
  progression-free survival is defined as the time from enrollment to the date of first document disease progression or death from any cause

SECONDARY OUTCOMES:
adverse event(AE) | Time Frame: approximately 36 months
  adverse event according to NCI CTCAE V4.0
overall survival (OS) | Time Frame: approximately over 3-5 years
  overall survival is defined as the time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No